CLINICAL TRIAL: NCT06652217
Title: Analysis of Occlusal Force Distribution in Digital and Conventional Occlusal Splint (Randomized Clinical Trial)
Brief Title: Analysis of Occlusal Force Distribution in Digital and Conventional Occlusal Splint
Acronym: splint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fatma hussein abd elmonem, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2497; ethics comittee (Other: 2497)
Record Dates: First submitted 2024-10-11; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the statistatian
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digitally manufactured occlusal splint (Experimental): digitally manfactured occlusal splint using intra oral scanner and jaw traccking device for data acqusition and 3d printing for manfacturing of the device
  Interventions: Device: Digitally manufactured occlusal splint.
- conventionally manufactured occlusal splint (Active Comparator): the occlusal device will be manufactured conventionally using impression and and anterior deprogramer with bite registeration material for data aquesition and usual construction method using clear acrylic.
  Interventions: Device: conventionally manufactured occlusal splint

INTERVENTIONS:
Device: Digitally manufactured occlusal splint. — digitally manfactured occlusal splint using intra oral scanner and jaw traccking device for data acqusition and 3d printing for manfacturing of the device
  Arms: Digitally manufactured occlusal splint
Device: conventionally manufactured occlusal splint — the occlusal device will be manufactured conventionally using impression and and anterior deprogramer with bite registeration material for data aquesition and usual construction method using clear acrylic.
  Arms: conventionally manufactured occlusal splint

SUMMARY:
Each eligible patient will be randomly into one of two groups:

Group A: The digital splint group, digital splint will be constructed to each patient.

Group B: The conventional splint group, conventional splint will be constructed to each patient.

* For both groups, thorough clinical examination, scaling and root-planning will be done. Patient will receive a motivational oral hygiene program with detailed explanation regarding the study process and outcome expectations.
* A precise history and clinical examination will be done by (F.M) under supervision of Dr S.G.

The digital splint construction method:

* First, complete arch intraoral digital scans of the maxillary and mandibular arches will be performed using the intra oral scanner following the scanning protocol recommended by the manufacturer.
* For inter maxillary relation recording using optical jaw tracking device, step-by-step procedure for tracking and recording the maxillomandibular relationship and mandibular motion by using an optical jaw tracking system will be illustrated to the patient.
* The occlusal device will be designed using a CAD software program.
* The occlusal device will be printed using a 3D printer
* The occlusal device will be finished and polished manually.

The conventional splint construction method:

* The first step is making an impression using a quick-setting addition polyvinyl siloxane impression material. A stone model will be obtained after pouring the impression using extra-hard dental stone.
* In the second visit a face bow transfer and a centric relation record will be utilized to mount the casts on a semi adjustable articulator.
* For centric relation recording, a jig will be made with an incisal plateau from modeling plastic impression compound and the jig will be inserted between the central incisors. To measure centric relation as precisely as possible (by avoiding translational movement in the temporomandibular joint),
* The jig will be adjusted with a scalpel to create a distance of no more than 2 mm between the maxillary and mandibular arches. Then the relation will be recorded using a fast-setting polyvinyl siloxane occlusal registration material. The occlusal registrations will be trimmed to the buccal cusp tips to be transferred accurately to the articulator without interference.
* After mounting of the centric relation the protrusive record will be taken and the horizontal condylar angle will be adjusted accordingly.
* The device will be fabricated from clear prosthetic resin. Production followed a standardized protocol with a minimum inter maxillary thickness of 1.5 mm and a buccal extension to 1 mm below the survey line.
* The device will be finished and occlusion will be adjusted on the articulator. outcomes assessment:

  1. Occlusal force distribution will be measured using osslusosense.
  2. Cost effectiveness will be assessed using the following equation(CE ratio = C/E).

ELIGIBILITY:
Inclusion Criteria:• Age range from 20 to 60 years old.

* Medically healthy patients.
* Patients with signs (as teeth attrition, muscles hypertrophy, and increased muscles activity) and symptoms (as muscles pain, headache, patient reporting) of bruxism for the last 6 months with no condylar or disc attrition.
* Fully dentate with presence of first molar in both arches
* Patients with good oral hygiene.
* Absence of any intra-oral pathological condition. Exclusion Criteria:• Patients with a history of psychosomatic disease.
* Patients with addiction to alcohol, drugs, or analgesics.
* Pregnant patients.
* Patients with malignant disease.
* Acute events such as trauma or inflammation.
* Bisphosphonate therapy within the last 5 years.
* Removable dental prostheses.
* Known hypersensitivity to materials.
* Extensive temporomandibular disorder that renders the stabilizing splints not to be the treatment of choice.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
occlusal force distribution | the outcome will be measured immediately after the device insertion
  the distribution of force between right and left side will be assessed using occlusosense device

SECONDARY OUTCOMES:
cost effectiveness | the outcome will be measured immediately after the device insertion
  the cost effectiveness will be measured using the following equation (CE ratio = C/E)

IPD SHARING:
Plan to Share IPD: No
iam not going to share the IPD for privacy and security of the informations